CLINICAL TRIAL: NCT02204397
Title: A Single-center, Open-Label, Exploratory Study to Assess the Tolerability and Safety of the Addition of Ustekinumab to INGAP Peptide for 12 Weeks in Adult Patients With Type 1 Diabetes Mellitus
Brief Title: Study of Tolerability and Safety of Adding Ustekinumab to INGAP Peptide for 12 Weeks in Adult Patients With TD1 Melitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Lawrence Rosenberg, Executive Director, Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JewishGH
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes mellitus; INGAP; Ustekinumab
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — INGAP peptide; Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- INGAP Peptide, Ustekinumab (Experimental): INGAP Peptide, Ustekinumab subcutaneous
  Interventions: Drug: INGAP Peptide, Ustekinumab

INTERVENTIONS:
Drug: INGAP Peptide, Ustekinumab
  Other Names: INGAP Peptide; Ustekinumab (Stelara)

SUMMARY:
A proof-of-concept for safety and preliminary clinical efficacy of a combined regimen of INGAP-P for β-cell regeneration and ustekinumab for IL-12-23 autoimmune modulation in patients with established T1DM.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the safety and tolerability of 12 weeks of subcutaneous (SC) daily administration of INGAP-P (600 mg SC once a day in three separate injection sites) with ustekinumab (two single injections of 45 mg SC, one as pretreatment two weeks before INGAP-P treatment begins and the second one after 2 weeks of INGAP-P treatment) in adult patients with established type 1 diabetes mellitus (T1DM). Safety will be evaluated by assessing local tolerability, recording incidence of hypoglycemia, performing safety laboratory measures at frequent intervals, and following subjects very closely for any adverse events (AEs).

Secondary objectives of this study are to generate preliminary data on the efficacy of INGAP-P and ustekinumab in adult patients with established T1DM, specifically by change from baseline to Week 12 in: 1) Maximal C-peptide (Cmax) during mixed meal test (MMT) and glucagon stimulated test (GST); 2) C-peptide release (AUC) during MMT and GST; 3) Fasting C-peptide; 4) Fasting glucose (before breakfast and after at least 8 hours of fasting); 5) Longer term glycemic control as reflected by glycosylated hemoglobin (HbA1c) and 1,5-anhydroglucitol (1,5-AG); and, 6) Total daily insulin dose relative to body weight.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients between the ages of 19 and 40 years old, inclusive, with a history of T1DM for >2 years and ≤20 years;
2. Female patients will not be breast-feeding during the study or within at least seven days after the study is completed;
3. Receiving multiple daily insulin injections or insulin pump therapy for >2 years;
4. Body mass index (BMI) ≤32 kg/m2 and total body weight <100 kg;
5. HbA1c ≤8.2%,
6. Fasting C-peptide levels >0.1 ng/mL and <1.0 ng/mL;
7. CBC and platelet counts must be within normal limits, and specifically, the total absolute neutrophil count must not be <1500/μL;
8. Willing to sign the study informed consent document;
9. In good general health with no infections, active tuberculosis (TB), late severe complications, or concomitant medical conditions that would influence the outcome of the trial, at the discretion of the Investigator and the Sponsor;
10. If treated with angiotensin-converting enzymes/angiotensin II receptor blockers (ACE/ARB), the doses should be unchanged for a month prior to enrollment;
11. Females of child bearing potential must have a negative urine pregnancy test on Day 0 prior to dispensing drug and should additionally fulfill one of the following criteria:

    * Willing to use oral, implantable, transdermal, or injectable contraceptives for 21 days prior to the first dose and until 28 days after the last dose; or,
    * Willing to use another reliable means of contraception approved by the Investigator (intrauterine device, female condom, diaphragm with spermicide, cervical cap, use of condom by sexual partner, or a sterile sexual partner) from Screening until after the last blood sample (at Week 16).

Exclusion Criteria:

1. Total daily insulin dosage exceeding 1.0 U/kg/day or a change in total daily insulin dose level of more than 50% (increase or decrease) within the past 3 months;
2. Treatment with any diabetes medication other than insulin;
3. A score of 4 or more restricted responses on the Clarke Hypoglycemia Awareness Survey;
4. Systolic or diastolic blood pressure >180 mmHg or >110 mmHg, respectively;
5. Clinical worsening of retinopathy or neuropathy in the previous 3 months;
6. Clinical worsening of nephropathy in the previous 3 months, or serum creatinine exceeding 2.0 mg/dL,;
7. History or presence of acute or chronic pancreatitis, including a serum amylase level >1.5 times the upper limit of normal (ULN) or a serum lipase level >2 times ULN;
8. Active infections at screening and during the study;
9. History of asthma;
10. History of TB;
11. Administration of bacille Calmette-Guérin (BCG) vaccine for TB during the one year before the Screening Visit or one year after the last dose of ustekinumab;
12. A history or presence of any illness, disease, or condition (including cancer) that could impact patient safety or evaluability of drug effect, in the Investigator"s opinion;
13. An episode of severe hypoglycemia (change in mental status requiring assistance) during the previous 30 days;
14. An episode of acute glycemic decompensation with associated hyperosmolar non-ketotic state or diabetic ketoacidosis during the past 6 months;
15. A serum aspartate aminotransferase (AST), alanine aminotransferase (ALT), or total bilirubin level >2 times ULN;
16. Received any investigational product within 30 days of admission into this study or had any prior or existing exposure to INGAP-P, glucagon-like peptides (GLP-1, GLP-2, or analogs), ustekinumab, or TNF blocking agents (Patients that participated in the placebo group of previous INGAP-P study E-201 are not excluded from this study.);
17. Known hypersensitivity to INGAP-P or any excipient used in the formulation;
18. Known hypersensitivity to ustekinumab or any components of the product;
19. Concurrent or planned participation in any other clinical study during the conduct of this study;
20. Positive urine test for cocaine, opiates, amphetamines, or cannabinoids;
21. Inability to fill out and maintain a daily diary during the screening period prior to dosing;
22. Human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C seropositivity in blood sample taken during screening.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2015-11; Primary Completion 2017-03-08 (Actual); Study Completion 2017-03-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 6 months
  The tolerability of injections and general safety will be assessed on the basis of patient recorded diaries, assessments of cutaneous injection sites during clinic visits, clinical observations, severity of AEs recorded by the Medical Dictionary for Regulatory Activities (MedDRA), measurement of vital signs, physical examinations, electrocardiograms (ECGs), and clinical laboratory evaluations.

SECONDARY OUTCOMES:
Composite C-Peptide efficacy according to specific parameters | 6 months
  Composite secondary objectives of this study are to generate preliminary data on the efficacy of INGAP-P and ustekinumab in adult patients with established T1DM, specifically by change from baseline to Week 12-13 in:
  * Maximal C-peptide (Cmax) during mixed meal test (MMT) and glucagon stimulated test (GST);
  * C-peptide release (AUC) during MMT and GST;
  * Fasting C-peptide;
  * Fasting glucose (before breakfast and after at least 8 hours of fasting);
  * Longer term glycemic control as reflected by glycosylated hemoglobin (HbA1c)

CONTACTS AND LOCATIONS:
Overall Officials: George Tsoukas, MD, Principal Investigator — Department of Endocrinology and Metabolism, Montreal General Hospital
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing is still under review and will be determined at a later date